CLINICAL TRIAL: NCT04860557
Title: Comparison of the Dual Task, Cognitive Skills and Physical Activity With Problematic Game Players and Control Subjects
Status: Completed | Type: Observational
Sponsor: Cagtay Maden (Other)
Responsible Party: Sponsor-Investigator, Cagtay Maden, research assistant,physiotherapist, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Other Study IDs: 2019/112
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Problematic Video Gaming; Cognitive Skill; Dual Task; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- problematic video game player
  Interventions: Other: cognitive skill, dual task and physical activity assessment
- control subjects
  Interventions: Other: cognitive skill, dual task and physical activity assessment

INTERVENTIONS:
Other: cognitive skill, dual task and physical activity assessment — Montreal Cognitive Assessment Test, Trail Making Test (TMT) A & B sections and Stroop test for cognitive ability assessment, 10 meter walking test (single-double task) for dual task, Time up and Go test (single-double task), physical International Physical Activity Questionnaire was used for activity and The Exercise Benefit / Barriers Scale was used for exercise perception.

SUMMARY:
This study was conducted to compare the cognitive skills, dual-task and physical activity status of individuals who play problem video games and healthy individuals, and to determine how much these skills are affected. The cognitive skills of individuals with video game playing problems and the control group were evaluated with the Montreal Cognitive Assessment Test, the Trail Making Test A & B sections, and the Stroop test. I evaluated dual tasks with 10-meter walking test (single-double task) and Time Up and Go Test (single-double task). Physical activity levels were evaluated by International Physical Active Questionnaire. The average cognitive skills, dual tasks, and physical activity levels of the individuals in both groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* DSM V (Diagnostic and Statistical Manual of Mental Disorders, revision 5) Internet Gaming Disorder (IOOB) Diagnostic criteria: Providing 5 out of 9 items
* No communication barrier
* To volunteer to participate in research
* Be playing games at least 2 hours a day in the last year

Exclusion Criteria:

* 3 days a week to be doing any sports
* Having a chronic illness
* Psychological disease diagnosis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students in Hasan Kalyoncu University
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 1 days
  It was used to evaluate the physical activities of individuals in the last week. It was also used to assess individuals' sedentary time.
The Exercise Benefits/Barriers Scale | 1 day
  This scale is used to measure exercise benefit perception. a high score indicates the presence of positive exercise perception. High scores on this scale indicate that the perception of obstacles to exercise is at the forefront.
Montreal Cognitive Assessment Test | 1 day
  Montreal Cognitive Assessment (MoCA) was developed as a rapid screening test for mild cognitive impairment.
Trail Making Test (TMT) A & B sections | 1 day
  It is one of the neuropsychological tests widely used all over the world. TMT is a test that requires visual-spatial processing and motor skills, which measures executive functions such as working memory, complex attention, planning, and set changes.
Stroop Test | 1 day
  It is a test that measures the ability to inhibition of inappropriate response in executive functions. It is a test that shows frontal functions that measures attention under a disruptive effect and evaluates to suppress inappropriate automatic responses.
10 meter walking test | 1 day
  the 10-meter walking test, subjects are walked at their own normal speed and the walking time is measured with a stopwatch and recorded in m / sec. In the beginning, the 2-meter assembling phase is accepted as the 2-meter deceleration phase at the end of the walk, and measurement is made on a 14-meter-long track. In our study, normal walking speed and dual walking speed were measured and recorded separately, accompanied by dual tasks. In the evaluation of dual walking speed, individuals were asked to count animal names starting with the letter "K" and walking speed was recorded.
Timed Up & Go (TUG) test | 1 day
  Timed Up & Go (TUG) test was used to evaluate functional mobility. Patients are asked to get up from the chair they are sitting in, walk 3 meters, turn back and sit on the chair again. Again, to evaluate the dual test, say words starting with the letter "N", the test is repeated and the time is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Universty, Gaziantep, Şahinbey, Turkey (Türkiye)